CLINICAL TRIAL: NCT04718649
Title: Effectiveness and Safety of Celecoxib (Celebrex 200 mg) Combined With Joins in the Treatment of Degenerative Knee Osteoarthritis: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KC20MISV0634
Record Dates: First submitted 2021-01-05; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Celebrex; Joins
MeSH Terms: conditions — Osteoarthritis | interventions — Celecoxib; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celebrex + Joins (Experimental): The experimental group will receive 12 weeks of Celebrex 200mg tab (taken once a day) and Joins (taken 3 times a day) at the clinical pharmacy at the first visit, and will be prescribed only Joins (taken 3 times a day) at week 12. They will only take Joins for another 24 weeks until the 36th week.
  The subject's oral medication is received at the clinical pharmacy twice at the time of first visit and at week 12. The follow-up period of the study will be 36 weeks.
  Interventions: Drug: Celebrex with Joins or not
- Celebrex + Placebo (Placebo Comparator): The control group will receive 12 weeks of Celebrex 200mg tab (taken once a day) and placebo (taken 3 times a day) at the clinical pharmacy at the first visit, and will be prescribed only placebo (taken 3 times a day) at week 12. They will only take Joins placebo for another 24 weeks until the 36th week.
  The subject's oral medication is received at the clinical pharmacy twice at the time of first visit and at week 12. The follow-up period of the study will be 36 weeks.
  Interventions: Drug: Celebrex with Joins or not

INTERVENTIONS:
Drug: Celebrex with Joins or not — The enrolled patienst will be divided into the group taking celecoxib 200mg with Joins tab together and the group taking celecoxib 200mg with Joins placebo in the same probability of 2:1 according to the randomization table at the first outpatient visit. Among the co-researchers, one researcher who is in charge of patient assignment will create a randomization table through computer generated randomization. And this researcher who is charge of the patient assignment will not intervene in any other process of this study, and only participates in the task of selecting the assigned group using random checks. The evaluation will be evaluated by an researcher who is not aware of the patient allocation according to the randomization table among researchers participating in the clinical study

SUMMARY:
Osteoarthritis of the knee joint causes pain, stiffness, and restriction of joint movement in the knee joint due to degeneration of the knee cartilage. The purpose of osteoarthritis treatment is to improve the joint pain and prevent further damage to the joint. Selective Cox-2 inhibitors are the most commonly used nonsteroid anti-inflammatory drugs(NSAIDs) for the treatment of osteoarthritis of the knee joint. However, the safety of selective Cox-2 inhibitors is still controversial. Although these NSAIDs are effective in reducing pain and inflammation, they cannot be called a fundamental treatment for knee arthritis. Accordingly, interest in SYSADOA (Symptomatic Slow-acting Drugs for Osteoarthritis) is gradually increasing.

Joins is a herbal anti-arthritic drug that has various physiological activities and a new concept of osteoarthritis treatment. It has anti-inflammatory, analgesic and joint cartilage protection effects as well as fundamental treatment. Joins is used to improve articular cartilage metabolism, can delay the progression of degenerative arthritis in the knee and compensate for the disadvantages of Selective Cox-2 inhibitors. However, when the selective Cox-2 inhibitor and Joins tablet are used alone, the therapeutic effect on knee degenerative arthritis may be limited. The purpose of this study is to investigate the therapeutic effect and safety of joining together with celecoxib for degenerative arthritis of the knee joint, and to determine the degree of analgesic and anti-inflammatory effects of the combination therapy.

DETAILED DESCRIPTION:
The Investigators will conduct research to patients with outpatient treatment for osteoarthritis of the knee joint, pain control will be performed using the same pain control technique that is generally applied to patients with osteoarthritis of the knee joint.

The enrolled patienst will be divided into the group taking celecoxib 200mg with Joins tab together and the group taking celecoxib 200mg with Joins placebo in the same probability of 2:1 according to the randomization table at the first outpatient visit. Among the co-researchers, one researcher who is in charge of patient assignment will create a randomization table through computer generated randomization. And this researcher who is charge of the patient assignment will not intervene in any other process of this study, and only participates in the task of selecting the assigned group using random checks. The evaluation will be evaluated by an researcher who is not aware of the patient allocation according to the randomization table among researchers participating in the clinical study. Such a study plan will be fully explained to the patient in the process of seeking consent for the study before discharge, as it is recorded in detail in the subject description, and only patients who have obtained consent for this will be the subject of the study.

Subjects assigned through randomization are prescribed and taken through the clinical pharmacy. Considering that Joins tab is a sustained-acting drug, the study is divided into Celebrex + Joins placebo group and Celebrex + Joins tab group for up to 12 weeks, and only Joins placeb and Joins are taken for weeks 12th week to 36th week except for celebrex. The total period of the study should be 36 weeks. In the case of the rescue drug, 650mg of Tylenol sustained-release tablet (acetaminophen) in both groups can be taken up to 3 tablets per day, and up to 36 weeks of taking the test drug. Patients should follow the approved usage and dosage, and taking relief drug is prohibited within 1 day before the regular visit. Relief drugs will be prescribed at baseline and from subsequent visits, if necessary, according to the judgment of the investigator.

At the first visit, at 4 weeks, 12 weeks, 24 weeks, 36 weeks, the degree of pain will be measured using the VAS pain scale, and additional pain scale using the WOMAC pain scale, Brief pain inventory (BPI), and SF-36 score.

Knee X-rays will be taken at each outpatient visit as the knee degenerative osteoarthritis patients are measured to check joint space width (JSW) and Kellgren-Lawrence grade to objectively evaluate the effectiveness and stability of the medication effect.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 50
* Patients undergoing outpatient treatment in orthopedic surgery for osteoarthritis of the knee joint
* Patients diagnosed with Kellgren-Lawrence grade II or III osteoarthritis of the knee by imaging examination
* Patients with a pain VAS scale of 4 or more out of 10 with a pain in the knee joint during daily activities on flat ground
* Patients confirmed by the examiner for no abnormal results in blood tests, etc.
* Patients who are willing or able to follow doctor's instructions, including joint exercises
* Patients not participating in other clinical trials
* Patients who have received sufficient explanation for this clinical trial and agreed to participate

Exclusion Criteria:

* Patients with secondary knee osteoarthritis
* Patients with hypersensitivity reactions and serious side effects to Celebrex or Joins
* Patients with inflammatory arthritis or crystalline arthritis
* Local infection to the lower extremities of the pain area, sepsis, or previous neurological abnormalities.
* Patients who underwent meniscus surgery on the knee joint in the painful area
* Patients who underwent total knee arthroplasty within 180 days of the knee joint opposite the pain area
* If there is construction or deformation of the knee joint in the pain area
* Patients with serious heart-related diseases such as cardiac arrest, a history of cerebral infarction, or ischemic heart disease
* Hemoglobin A1c level >8% of patients not managed by diabetes
* Patients with high blood pressure with poor blood pressure control (Systolic Blood Pressure of> 150 mmHg or Diastolic Blood Pressure> 95 mmHg)
* Patients taking PPI drugs for recurrent upper gastrointestinal ulcer or inflammatory bowel disease (such as Crohn's disease or ulcerative colitis)
* Patients with abnormal liver function (ALT)> 2.0 times the upper limit of normal (ULN) or blood urea nitrogen (BUN) or serum creatinine> 2.0 times ULN)
* Patients who took excessive narcotic analgesics for pain in the affected area before the clinical trial
* Patients scheduled for surgery during the clinical trial period
* Patients who received intraarticular injection treatment into the painful area of the knee within 3 months prior to the first visit
* Patients who received systemic steroid treatment within 3 months prior to their first visit
* Pregnant or lactating women

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC(Western Ontario and McMaster University Arthritis Index ) pain scale | changes of the WOMAC score from the first day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | First day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment
Brief pain inventory (BPI) | First day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment
SF-36 score | First day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment
Serum Biomarker | First day of enrollment, 12th week after enrollment, 36th week after enrollment
  CTX-1, CTX-2. COMP, HA, NTX-1
X-ray | First day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment
  joint space width, Kellgren-Lawrence grade
Adverse event | First day of enrollment, 4th week after enrollment, 12th week after enrollment, 24th week after enrollment, 36th week after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- the Catholic Univerisity of Korea Seoul St Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No